CLINICAL TRIAL: NCT02185105
Title: Clinical Validation of Biofinity Toric MTO (Made To Order) Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CV-14-04
Record Dates: First submitted 2014-07-07; First posted 2014-07-09 (Estimated); Results first posted 2017-01-02 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- comfilcon A MTO (Experimental): Subjects will be randomized to receive either the Test or Control lens as a matched pair at each visit per a predetermined randomization schedule.
  Interventions: Device: comfilcon A
- comfilcon A (Active Comparator): Subjects will be randomized to receive either the Test or Control lens as a matched pair at each visit per a predetermined randomization schedule.
  Interventions: Device: comfilcon A MTO

INTERVENTIONS:
Device: comfilcon A MTO — Randomized to a test lens in one eye and control lens in the other as a matched pair.
  Other Names: Biofinity Toric MTO
  Arms: comfilcon A
Device: comfilcon A — Randomized to a test lens in one eye and control lens in the other as a matched pair.
  Other Names: Biofinity Toric
  Arms: comfilcon A MTO

SUMMARY:
The study hypothesis is there is no difference in the clinical performance between the test and control lenses, in particular in lens stability, toric mislocation, comfort ratings and anterior segment ocular health findings.

DETAILED DESCRIPTION:
Evaluate the clinical performance of Biofinity toric MTO lenses against current commercial Biofinity toric lenses over 6 hours of lens wear.

ELIGIBILITY:
Inclusion Criteria:

* Has had a self-reported oculo-visual examination in the last two years.
* Is at least 18 years of age and has full legal capacity to volunteer.
* Has read and understood the information consent letter.
* Is willing and able to follow instructions and maintain the appointment schedule.
* Is correctable to a visual acuity of 20/40 or better (in each eye) with their habitual vision correction or 20/20 best-corrected.
* Currently wears soft contact lenses.
* Has clear corneas and no active ocular disease.
* Has not worn lenses for at least 12 hours before the examination

Exclusion Criteria:

* Has never worn contact lenses before.
* Has any systemic disease affecting ocular health.
* Is using any systemic or topical medications that will affect ocular health.
* Has any ocular pathology or severe insufficiency of lacrimal secretion (moderate to severe dry eyes) that would affect the wearing of contact lenses.
* Has persistent, clinically significant corneal or conjunctival staining using sodium fluorescein dye.
* Has any clinically significant lid or conjunctival abnormalities, active neovascularization or any central corneal scars.
* Is aphakic.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pete S Kollbaum, O.D., Principal Investigator — Indiana University
Locations (1):
- CORL, Indiana University, Bloomington, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Comfilcon A XR Toric (Extended Range) / Comfilcon A Toric: Subjects were randomized to receive either the Test or Control lens as a matched pair at each visit per a predetermined randomization schedule.
  comfilcon A: Randomized to a test lens in one eye and control lens in the other as a matched pair.
Period: Overall Study
Arm/Group | Comfilcon A XR Toric (Extended Range) / Comfilcon A Toric
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Comfilcon A XR Toric (Extended Range) / Comfilcon A Toric
Number analyzed (Participants) | 30
Age, Customized [Number; unit: participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Lens Surface Assessment of Study Lenses - Surface Wettability
Description: Investigator's objective assessment of lens surface wettability at 15min and 6hrs. Scale (0-4; 0=non-wetting, 4=Excellent)
Time Frame: 15min & 6hrs
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Comfilcon A XR (Extended Range) Toric: Subjects were randomized to receive either the Test or Control lens as a matched pair at each visit per a predetermined randomization schedule.
  comfilcon A: Randomized to a test lens in one eye and control lens in the other as a matched pair.
- Comfilcon A Toric: Subjects will be randomized to receive either the Test or Control lens as a matched pair at each visit per a predetermined randomization schedule.
  comfilcon A XR: Randomized to a test lens in one eye and control lens in the other as a matched pair.
Arm/Group | Comfilcon A XR (Extended Range) Toric | Comfilcon A Toric
Number analyzed (Participants) | 30 | 30
units on a scale
  15 minutes | 3.4 (0.3) | 3.4 (0.2)
  6 hours | 3.4 (0.4) | 3.4 (0.4)

2. Primary Outcome: Lens Surface Assessment of Study Lenses - Deposits
Description: Investigator's objective assessment of lens surface deposition at 15min and 6hrs. Graded on the appearance of lens surface by slit lamp. Rated on a scale (0-4; 0=no deposits, 4=deposits ≥0.5mm or film > 75% of surface)
Time Frame: 15min & 6hrs
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Comfilcon A XR Toric (Extended Range): Subjects were randomized to receive either the Test or Control lens as a matched pair at each visit per a predetermined randomization schedule.
  comfilcon A: Randomized to a test lens in one eye and control lens in the other as a matched pair.
Arm/Group | Comfilcon A XR Toric (Extended Range) | Comfilcon A Toric
Number analyzed (Participants) | 30 | 30
units on a scale
  15 minutes | 0.00 (0.00) | 0.00 (0.00)
  6 hours | 0.03 (0.18) | 0.00 (0.00)

3. Primary Outcome: Lens Surface Assessment of Study Lenses - Surface Acceptance
Description: Investigator's objective assessment of surface acceptance at 15min and 6hrs. Rated on a scale (0-4; 0=very poor, 4=excellent)
Time Frame: 15min & 6hrs
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A XR Toric (Extended Range) | Comfilcon A Toric
Number analyzed (Participants) | 30 | 30
units on a scale
  15 minutes | 3.4 (0.4) | 3.4 (0.4)
  6 hours | 3.4 (0.5) | 3.4 (0.5)

4. Primary Outcome: Subjective Rating For Comfort - Comfort Since Last Visit
Description: Participant's subjective rating of comfort now of study lenses. Surveyed at 15min, 3hr, and 6hr. Scale (0-100; 0=cannot be worn, causes pain, 100=cannot be felt ever)
Time Frame: 15min, 3hrs, 6hrs
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A XR Toric (Extended Range) | Comfilcon A Toric
Number analyzed (Participants) | 30 | 30
units on a scale
  15 minutes | 88 (11) | 90 (10)
  3 hours | 84 (17) | 87 (12)
  6 hours | 84 (15) | 88 (11)

5. Primary Outcome: Subjective Rating For Comfort Preference
Description: Participant's subjective rating of comfort preference of study lenses. Scale: (Strongly Prefer Right lens - Strongly Prefer Left Lens)
Time Frame: 1min, 15min, 3hrs, 6hrs
Measure: Number; unit: percentage of subjects
Arm/Group | Comfilcon A XR Toric (Extended Range) | Comfilcon A Toric | No Preference
Number analyzed (Participants) | 30 | 30 | 30
percentage of subjects
  1 minute | 23 | 47 | 30
  15 minutes | 23 | 47 | 30
  3 hours | 17 | 30 | 53
  6 hours | 20 | 37 | 43

6. Primary Outcome: Subjective Rating For Handling - Insertion
Description: Participant's subjective rating for ease of insertion of the study lenses. Scale (0-100; 0=could not place lens on eye;100=always easy to place lens on eye)
Time Frame: 1 min
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A XR Toric (Extended Range) | Comfilcon A Toric
Number analyzed (Participants) | 30 | 30
units on a scale | 95 (7) | 95 (7)

7. Primary Outcome: Subjective Rating For Handling - Removal
Description: Participant's subjective rating for ease of removal of study lenses. Scale (0-100; 0=could not remove lens from eye;100=always easy to place remove from eye)
Time Frame: 1 min
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A XR Toric (Extended Range) | Comfilcon A Toric
Number analyzed (Participants) | 30 | 30
units on a scale | 63 (38) | 74 (30)

8. Primary Outcome: Investigator's Assessment of Stability
Description: Investigator's assessment of the study lenses overall stability difference measured from 0-180 degrees, 0=very good stability, 180=very bad stability.
Time Frame: 15min & 6hrs
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Comfilcon A XR Toric (Extended Range) | Comfilcon A Toric
Number analyzed (Participants) | 30 | 30
degrees
  15 minutes | 3 (4) | 3 (3)
  6 hours | 3 (3) | 4 (7)

9. Primary Outcome: General Lens Fit - Fit Acceptance
Description: Investigator's assessment for fit acceptance of study lenses. Scale: 0-4 (0=Should not be worn; 4=Perfect)
Time Frame: 15min & 6hrs
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A XR Toric (Extended Range) | Comfilcon A Toric
Number analyzed (Participants) | 30 | 30
units on a scale
  15 minutes | 3.4 (0.2) | 3.4 (0.2)
  6 hours | 3.4 (0.2) | 3.4 (0.2)

10. Primary Outcome: Lens Fitting - Rotation/Mislocation
Description: Investigator's observed the rotation/mislocation (toric mark) of study lenses from the desired 6 o'clock position following temp rotation 30 degrees, 10 blinks; rotation toward desired 6 o'clock position=(+); rotation away from desired 6 o'clock position=(-).
Time Frame: Baseline, 15min & 6hrs
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Comfilcon A XR Toric (Extended Range) | Comfilcon A Toric
Number analyzed (Participants) | 30 | 30
degrees
  Baseline | 1 (5) | 3 (9)
  15 minutes | 1 (6) | 1 (7)
  6 hours | 2 (5) | -1 (7)

11. Primary Outcome: Anterior Ocular Health - Corneal Staining (Central)
Description: Corneal staining (central) for comfilcon (A) toric and comfilcon (A) toric XR lenses assessed at baseline and 6 hours. (Scale 0-4, 0=No staining; 4= >45% of area)
Time Frame: baseline & 6hrs
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comflicon A XR Toric (Extended Range) | Comfilcon A Toric
Number analyzed (Participants) | 30 | 30
units on a scale
  Baseline | 0.02 (0.09) | 0.02 (0.09)
  6 hours | 0.00 (0.00) | 0.00 (0.00)

12. Primary Outcome: Anterior Ocular Health - Corneal Staining (Nasal)
Description: Corneal staining (nasal) for comfilcon (A) toric and comfilcon (A) toric XR lenses assessed at baseline and 6 hours. (Scale 0-4, 0=No staining; 4= >45% of area)
Time Frame: baseline & 6hrs
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comflicon A XR Toric (Extended Range) | Comfilcon A Toric
Number analyzed (Participants) | 30 | 30
units on a scale
  Baseline | 0.02 (0.09) | 0.05 (0.20)
  6 hours | 0.00 (0.00) | 0.00 (0.00)

13. Primary Outcome: Anterior Ocular Health - Corneal Staining (Temporal)
Description: Corneal staining (temporal) for comfilcon (A) toric and comfilcon (A) toric XR lenses assessed at baseline and 6 hours. (Scale 0-4, 0=No staining; 4= >45% of area)
Time Frame: baseline & 6hrs
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comflicon A XR Toric (Extended Range) | Comfilcon A Toric
Number analyzed (Participants) | 30 | 30
units on a scale
  Baseline | 0.02 (0.09) | 0.05 (0.20)
  6 hours | 0.00 (0.00) | 0.00 (0.00)

14. Primary Outcome: Anterior Ocular Health - CornealStaining (Superior)
Description: Corneal staining (superior) for comfilcon (A) toric and comfilcon (A) toric XR lenses assessed at baseline and 6 hours. (Scale 0-4, 0=No staining; 4= >45% of area)
Time Frame: baseline & 6hrs
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comflicon A XR Toric (Extended Range) | Comfilcon A Toric
Number analyzed (Participants) | 30 | 30
units on a scale
  Baseline | 0.00 (0.00) | 0.03 (0.18)
  6 hours | 0.02 (0.09) | 0.00 (0.00)

15. Primary Outcome: Anterior Ocular Health - Corneal Staining (Inferior)
Description: Corneal staining (inferior) for comfilcon (A) toric and comfilcon (A) toric XR lenses assessed at baseline and 6 hours. (Scale 0-4, 0=No staining; 4= >45% of area)
Time Frame: baseline & 6hrs
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comflicon A XR Toric (Extended Range) | Comfilcon A Toric
Number analyzed (Participants) | 30 | 30
units on a scale
  Baseline | 0.12 (0.31) | 0.05 (0.20)
  6 hours | 0.13 (0.35) | 0.28 (0.45)

16. Primary Outcome: Anterior Ocular Health - Conjunctival Staining (Nasal)
Description: Conjunctival staining (nasal) for comfilcon (A) toric and comfilcon (A) toric XR lenses assessed at baseline and 6 hours. Scale: 0-4, (0=None; 4=Deep confluent).
Time Frame: baseline & 6hrs
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comflicon A XR Toric (Extended Range) | Comfilcon A Toric
Number analyzed (Participants) | 30 | 30
units on a scale
  Baseline | 0.20 (0.41) | 0.13 (0.35)
  6 hours | 0.20 (0.41) | 0.23 (0.43)

17. Primary Outcome: Anterior Ocular Health - Conjunctival Staining (Superior)
Description: Conjunctival staining (superior) for comfilcon (A) toric and comfilcon (A) toric XR lenses assessed at baseline and 6 hours. Scale: 0-4, (0=None; 4=Deep confluent).
Time Frame: baseline & 6hrs
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comflicon A XR Toric (Extended Range) | Comfilcon A Toric
Number analyzed (Participants) | 30 | 30
units on a scale
  Baseline | 0.00 (0.00) | 0.00 (0.00)
  6 hours | 0.00 (0.00) | 0.03 (0.18)

18. Primary Outcome: Anterior Ocular Health - Conjunctival Staining (Temporal)
Description: Conjunctival staining (temporal) for comfilcon (A) toric and comfilcon (A) toric XR lenses assessed at baseline and 6 hours. Scale: 0-4, (0=None; 4=Deep confluent).
Time Frame: baseline & 6hrs
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comflicon A XR Toric (Extended Range) | Comfilcon A Toric
Number analyzed (Participants) | 30 | 30
units on a scale
  Baseline | 0.07 (0.25) | 0.00 (0.00)
  6 hours | 0.07 (0.25) | 0.13 (0.35)

19. Primary Outcome: Anterior Ocular Health - Conjunctival Staining (Inferior)
Description: Conjunctival staining (inferior) for comfilcon (A) toric and comfilcon (A) toric XR lenses assessed at baseline and 6 hours. Scale: 0-4, (0=None; 4=Deep confluent).
Time Frame: baseline & 6hrs
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comflicon A XR Toric (Extended Range) | Comfilcon A Toric
Number analyzed (Participants) | 30 | 30
units on a scale
  Baseline | 0.03 (0.18) | 0.00 (0.00)
  6 hours | 0.10 (0.31) | 0.10 (0.31)

ADVERSE EVENTS:
Arm/Group | Comfilcon A MTO | Comfilcon A
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study.

There is an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

The investigators will not be permitted to publish or present at scientific meetings results obtained from the clinical study without prior written consent from the sponsor.